CLINICAL TRIAL: NCT01503827
Title: Whole Brain Radiotherapy Following Local Treatment of Intracranial Metastases of Melanoma - A Randomised Phase III Trial
Brief Title: Whole Brain Radiotherapy Following Local Treatment of Intracranial Metastases of Melanoma
Acronym: WBRTMel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Trans Tasman Radiation Oncology Group (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-07; ACTRN12607000512426 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2011-12-15; First posted 2012-01-04 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Melanoma
Keywords: Whole Brain Radiotherapy; Brain metastases; Melanoma; Stage IV Metastatic Melanoma; Neurocognitive function; Quality of life
MeSH Terms: conditions — Melanoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WBRT (Experimental): Patients will receive WBRT after local treatment. A minimum of 30 Gy in 10 fractions given as one fraction per day within 4 weeks of randomisation
  Interventions: Radiation: WBRT
- Observation (No Intervention): No Intervention

INTERVENTIONS:
Radiation: WBRT — A minimum of 30 Gy in 10 fractions given as one fraction per day within 4 weeks of randomisation
  Arms: WBRT

SUMMARY:
People with brain metastases from melanoma are offered different treatment options after local treatment of their brain metastases via surgery or stereotactic irradiation. Depending on the treating institution and the clinician involved a patient may or may not be offered whole brain radiotherapy (WBRT) after their brain metastases are excised or treated with stereotactic irradiation. This trial seeks to determine if WBRT reduces the spread of brain metastases and lengthens the time to recurrence. The trial also examines the effect of WBRT on quality of life and brain functions such as memory, speech and concentration. Participants will be randomised after local treatment of their brain metastases to either WBRT or observation. 220 people will be recruited from sites in Australia, Norway, the UK, the US and other international sites.

ELIGIBILITY:
Inclusion Criteria:

* 1-3 intracranial metastases on MRI from melanoma, locally treated with either surgical excision and/or stereotactic irradiation.
* Life expectancy of at least 6 months
* Aged 18 years or older
* WBRT must begin within 8 weeks of completion of localised treatment and within 4 weeks of randomisation
* Able to have an MRI brain scan with contrast. Estimated Glomerular Filtrate Rate (eGFR) is adequate at the discretion of the radiologist and capable of having gadolinium-containing contrast medium for MRI as per practice guidelines
* Complete localised treatment of all these metastases no more than 6 weeks prior to randomisation
* An Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less at randomisation
* CT scan of chest, abdomen and pelvis as a minimum prior to randomisation. Scans must be within 12 weeks of randomisation
* Serum Lactate Dehydrogenase (LDH) must be = or < 2 x upper limit of normal
* Able to provide written informed consent

Exclusion Criteria:

* Any untreated intracranial disease
* Any previous intracranial treatment (surgical excision and/or stereotactic irradiation treatment and/or WBRT) prior to this diagnosis of intracranial melanoma
* Evidence of leptomeningeal disease on pre-local treatment MRI scan
* Patients with prior cancers, except:

  * Those diagnosed more than five years ago with no evidence of disease recurrence within this time;
  * Successfully treated basal cell and squamous cell skin carcinoma;
  * Carcinoma in-situ of the cervix
* A medical or psychiatric condition that compromises ability to give informed consent or complete the protocol
* Positive urine pregnancy test for women of childbearing potential within a week of registration onto the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-10; Primary Completion 2017-09 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with distant intracranial failure as determined by magnetic resonance imaging (MRI) assessment | 12 months post randomisation

SECONDARY OUTCOMES:
Time to intracranial failure (local, distant and overall) as determined by MRI | Post randomisation to intracranial failure
Quality of life as measured by EORTC QLQ-C30 and BN-20 | At baseline and every 2 months post randomisation
Neurocognitive function as measured by Hopkins Verbal Learning Test, Controlled Oral Word Association Test, Trail Making Test Part A & B, Stroop - Colour and Word Test and Digit Span (Forwards and Backwards). | At baseline and every 2 months post randomisation
Overall survival | Post randomisation to death from any cause
Performance status as measured by ECOG | At baseline and every 2 months post randomisation
Incremental cost effectiveness ratio (ICER) | At 12 months from randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Fogarty, BSc, MBBS, Study Chair — Mater Hospital, St Vincent's Hospital, Melanoma Institue Australia
Locations (23):
- Australia (17):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Calvary Mater Hospital, Newcastle, New South Wales
  - Genesis Cancer Care - Gateshead, Newcastle, New South Wales
  - Melanoma Institute Australia / Royal Prince Alfred Hospital, North Sydney, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Darwin Hospital, NT Radiation Oncology, Darwin, Northern Territory
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Radiation Oncology Services - Mater Centre, South Brisbane, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Genesis Cancer Care - Tugun, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- The Norwegian Radium Hospital, Oslo, Norway
- United Kingdom (5):
  - Velindre Hospital, Whitchurch, Cardiff
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Churchill Hospital, Headington, Oxford
  - St. James University Hospital, Leeds
  - Norfolk & Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fogarty G, Morton RL, Vardy J, Nowak AK, Mandel C, Forder PM, Hong A, Hruby G, Burmeister B, Shivalingam B, Dhillon H, Thompson JF. Whole brain radiotherapy after local treatment of brain metastases in melanoma patients--a randomised phase III trial. BMC Cancer. 2011 Apr 17;11:142. doi: 10.1186/1471-2407-11-142. PMID 21496312
- [Derived] Bartula I, Tran AD, Nowak AK, Ahmed T, Morton RL, Burmeister BH, Dolven-Jacobsen K, Nobes J, Thompson JF, Fogarty GB, Lo SN, Hong AM. Longitudinal trajectory of quality of life for patients with melanoma brain metastases: A secondary analysis from a whole brain radiotherapy randomized clinical trial. Clin Transl Radiat Oncol. 2023 Feb 15;41:100597. doi: 10.1016/j.ctro.2023.100597. eCollection 2023 Jul. PMID 37441544
- [Derived] Hong AM, Fogarty GB, Dolven-Jacobsen K, Burmeister BH, Lo SN, Haydu LE, Vardy JL, Nowak AK, Dhillon HM, Ahmed T, Shivalingam B, Long GV, Menzies AM, Hruby G, Drummond KJ, Mandel C, Middleton MR, Reisse CH, Paton EJ, Steel V, Williams NC, Scolyer RA, Morton RL, Thompson JF. Adjuvant Whole-Brain Radiation Therapy Compared With Observation After Local Treatment of Melanoma Brain Metastases: A Multicenter, Randomized Phase III Trial. J Clin Oncol. 2019 Nov 20;37(33):3132-3141. doi: 10.1200/JCO.19.01414. Epub 2019 Sep 25. PMID 31553661
- [Derived] Lo SN, Hong AM, Haydu LE, Ahmed T, Paton EJ, Steel V, Hruby G, Tran A, Morton RL, Nowak AK, Vardy JL, Drummond KJ, Dhillon HM, Mandel C, Scolyer RA, Middleton MR, Burmeister BH, Thompson JF, Fogarty GB. Whole brain radiotherapy (WBRT) after local treatment of brain metastases in melanoma patients: Statistical Analysis Plan. Trials. 2019 Aug 5;20(1):477. doi: 10.1186/s13063-019-3555-5. PMID 31382986
- See also: Click here for more information about this study: Whole Brain Radiotherapy following local treatment of intracranial metastases of melanoma — http://anzmtg.org/trialdetails.aspx?trialno=5